CLINICAL TRIAL: NCT05722106
Title: Improving Adherence to COVID-19 Prevention Behaviours: Test of Persuasive Messages
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: REB21-0173
Record Dates: First submitted 2023-01-10; First posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Control - Info only (Experimental): Participants read a flyer containing the following message:
  The virus spreads mainly between people who are in close contact with one another. You can help prevent the spread of COVID-19. We can all do our part:
  * Avoid social gatherings.
  * Wear a mask when you go out.
  * Stay at least six feet away from people outside your household.
  * Wash your hands often with soap and water. These actions prevent the spread of COVID-19.
  Interventions: Behavioral: Persuasive Appeal
- Deontological (Experimental): Participants read a flyer containing the following message:
  The virus spreads mainly between people who are in close contact with one another. You can help prevent the spread of COVID-19. We can all do our part:
  * Avoid social gatherings.
  * Wear a mask when you go out.
  * Stay at least six feet away from people outside your household.
  * Wash your hands often with soap and water. We all need to do this, however difficult, because it is the right thing to do: it is our duty and responsibility to protect our families, friends, and fellow citizens.
  Interventions: Behavioral: Persuasive Appeal
- Empathy (Experimental): Participants read a flyer containing the following message:
  The sick, elderly, and immunocompromised need our help. We all have a choice. If we don't take the right actions, we risk the lives of others. But we can protect those most likely to be harmed. We can protect those who are vulnerable by taking simple steps:
  * Avoid social gatherings.
  * Wear a mask when you go out.
  * Stay at least six feet away from people outside your household.
  * Wash your hands often with soap and water. Take action to protect those who are vulnerable!
  Interventions: Behavioral: Persuasive Appeal
- Identifiable victim (Experimental): Participants read a flyer containing the following message:
  A few weeks ago, Sam was a healthy 26-year-old with no medical complications. The he suddenly came down with a bad cough and a feeling like he could not breath. He tested positive for COVID-19, and is now hospitalized, receiving oxygen from a ventilator, and fighting for his life. This could be any of us. Reduce the risk to yourself and other:
  * Avoid social gatherings.
  * Wear a mask when you go out.
  * Stay at least six feet away from people outside your household.
  * Wash your hands often with soap and water. If we take these actions, we can prevent more people from suffering the way Sam has.
  Interventions: Behavioral: Persuasive Appeal
- Goal proximity (Experimental): Participants read a flyer containing the following message:
  The recent development of safe and effective vaccines gives us great hope. We see the light at the end of the tunnel, but we are not quite there yet. Until a large proportion of the population is immunized, we must remain vigilant and double our efforts to prevent the spread of COVID-19.
  * Avoid social gatherings.
  * Wear a mask when you go out.
  * Stay at least six feet away from people outside your household.
  * Wash your hands often with soap and water. These actions prevent the spread of COVID-19.
  Interventions: Behavioral: Persuasive Appeal
- Reciprocity (Experimental): Participants read a flyer containing the following message:
  Doctors, nurses, and other healthcare workers are working around the clock, often risking their lives to care for patients with the coronavirus. Working long hours in highly infectious environments, many of them are falling ill. As our healthcare workers put their lives on the line, we can do our part:
  * Avoid social gatherings.
  * Wear a mask when you go out.
  * Stay at least six feet away from people outside your household.
  * Wash your hands often with soap and water. Our brave healthcare workers have sacrificed to help others. We should take action too.
  Interventions: Behavioral: Persuasive Appeal

INTERVENTIONS:
Behavioral: Persuasive Appeal — Persuasive appeals were manipulated using promotional flyers ostensibly distributed by the Public Health Agency of Canada.

SUMMARY:
The goal of this randomized online experiment was to test the effectiveness of using various persuasive appeals (deontological moral frame, empathy, identifiable victim, goal proximity, and reciprocity) at improving intentions to adhere to prevention behaviors.

Participants indicated their intentions to follow public health guidelines, saw one of six flyers featuring a persuasive appeal or no appeal, then rated their intentions a second time. Known correlates of attitudes toward public health measures were also measured.

DETAILED DESCRIPTION:
Adherence to non-pharmaceutical interventions (NPIs) for COVID-19, including physical distancing, masking, staying home while sick, and avoiding crowded indoor spaces remain critical for limiting the spread of COVID-19.

This study tests the effectiveness of using various persuasive appeals (deontological moral frame, empathy, identifiable victim, goal proximity, and reciprocity) at improving intentions to adhere to prevention behaviors.

A randomized online experiment using a representative sample of adult Canadian residents with respect to age, ethnicity, and province of residence was conducted between March 3-6, 2021. Participants indicated their intentions to follow public health guidelines, saw one of six flyers featuring a persuasive appeal or no appeal, then rated their intentions a second time. Known correlates of attitudes toward public health measures were also measured.

ELIGIBILITY:
Inclusion Criteria:

* Adult Canadian residents
* Target quotas for province of residence, age, gender, and ethnicity were set to obtain a demographically representative sample based on the 2016 census data

Exclusion Criteria:

* Province of residence, age, gender, and ethnicity once quotas are filled

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3746 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2021-03-06 (Actual); Study Completion 2021-03-06 (Actual)

PRIMARY OUTCOMES:
Change in intentions to engage in prevention behaviours | Same day
  Index variables for intentions to engage in prevention behaviors (pre- and post-treatment) were created by averaging across six items (1. Limit my physical contact with others when possible, 2. Completely avoid any unnecessary physical contact with others [e.g., hugging or handshakes], 3. Avoid crowded indoor spaces, 4. Wear a mask when I leave the house, 5. Wash my hands as much as possible, and 6. Stay home when mildly sick) measured on 100-point sliding scales (0 = Strongly disagree, 50 = Neither agree nor disagree, 100 = Strongly agree).

CONTACTS AND LOCATIONS:
Overall Officials: Mehdi Mourali, PhD, Principal Investigator — University of Calgary
Locations (1):
- Lucid Marketplace, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mourali M, Benham JL, Lang R, Fullerton MM, Boucher JC, Cornelson K, Oxoby RJ, Constantinescu C, Tang T, Marshall DA, Hu J. Persuasive Messages for Improving Adherence to COVID-19 Prevention Behaviors: Randomized Online Experiment. JMIR Hum Factors. 2023 Feb 13;10:e41328. doi: 10.2196/41328. PMID 36508732